CLINICAL TRIAL: NCT03566576
Title: Dose Climbing Trial of Anlotinib Plus Pemetrexed/Docetaxel in the Second-line Treatment of Advanced Gene Negative Non-squamous Non-small Cell Lung Cancer
Brief Title: Phase I Study of the Combination of Anlotinib With Pemetrexed or Docetaxel
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FujianCH110
Record Dates: First submitted 2018-05-29; First posted 2018-06-25 (Actual); Last update posted 2018-06-25 (Actual); Status verified 2018-05

CONDITIONS: Non-squamous Non-small Cell Lung Cancer
MeSH Terms: interventions — anlotinib; Pemetrexed; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anlotinib Plus Pemetrexed (Experimental): This study will include a sequential evaluation of 3 subjects per cohort. Cohort 1: Anlotinib 8mg per day and Pemetrexed. Cohort 2: Anlotinib 10mg per day and Pemetrexed. Cohort 3: Anlotinib 12mg per day and Pemetrexed.
  A dose limiting toxicity (DLT) event is defined as any of the following events:
  1. CTCAE Grade 4 event (ANC<1000/ul, body temperature≥38.5°C);
  2. Grade 3 non-hematologic toxicity (except for nausea and vomiting that could be improved with optimal supportive care, escalation of alkaline phosphatase) If a DLT is experienced in any cohort, the cohort will be expanded to 6 subjects. If 2 DLTs are experienced in any cohort, the dose escalation ceased. The MTD was defined as the dose having at most two out of six patients experience DLT.
  Interventions: Drug: Anlotinib; Drug: Pemetrexed
- Anlotinib Plus Docetaxel (Experimental): This study will include a sequential evaluation of 3 subjects per cohort. Cohort 1: Anlotinib 8mg per day and Pemetrexed. Cohort 2: Anlotinib 10mg per day and Pemetrexed. Cohort 3: Anlotinib 12mg per day and Pemetrexed.
  A dose limiting toxicity (DLT) event is defined as any of the following events:
  1. CTCAE Grade 4 event (ANC<1000/ul, body temperature≥38.5°C);
  2. Grade 3 non-hematologic toxicity (except for nausea and vomiting that could be improved with optimal supportive care, escalation of alkaline phosphatase) If a DLT is experienced in any cohort, the cohort will be expanded to 6 subjects. If 2 DLTs are experienced in any cohort, the dose escalation ceased. The MTD was defined as the dose having at most two out of six patients experience DLT.
  Interventions: Drug: Anlotinib; Drug: Docetaxel

INTERVENTIONS:
Drug: Anlotinib — Anlotinib 8mg p.o. qd in first cohort (3 subjects). 10mg p.o. qd in second cohort (3 subjects). 12mg p.o. qd in third cohort (3 subjects).
Drug: Pemetrexed — Pemetrexed 500mg/m2 as a 10-minute intravenous infusion on day 1 of a 21-day cycle.
  Arms: Anlotinib Plus Pemetrexed
Drug: Docetaxel — Docetaxel 60mg/m2 as a 10-minute intravenous infusion on day 1 of a 21-day cycle.
  Other Names: Taxotere
  Arms: Anlotinib Plus Docetaxel

SUMMARY:
The purpose of this clinical study is to evaluate the tolerability and toxicity of different dose of Anlotinib puls Pemetrexed/Docetaxel in Second-line Treatment of Advanced Gene Negative Non-squamous Non-small Cell Lung Cancer , to provide a reference of dosage for Phase II clinical trials

DETAILED DESCRIPTION:
This is a randomized, single -center study conducted in China to compare the tolerability and toxicity of different dose of Anlotinib Plus Pemetrexed / Docetaxel in patients of Advanced Gene Negative Non-squamous Non-small Cell Lung Cancer.From low dose group up to high dose group, each one had 3 patients at least.Primary group received anlotinib 8mg. The dose of Anlotinib would increase gradually until MTD.

Eligible patients will be randomized to arm A and arm B:

Arm A: Patients were instructed to take folic acid 400ug orally daily beginning 1 week before the first dose of pemetrexed and continuing daily until 3 weeks after the last dose of pemetrexed. A 1000ug B12 injection was administered intramuscularly approximately 1 week before the first dose of pemetrexed and was repeated approximately every 9 weeks until after discontinuation. All target volumes were instructed to take dexamethasone (4 mg orally twice daily the day before, the day of, and the day after pemetrexed) as a prophylactic measure against skin rash. Patients on the pemetrexed arm received 500mg/m2 pemetrexed as a 10-minute intravenous infusion on day 1 of a 21-day cycle and 8mg/10mg/12mg Anlotinib orally daily on day 1 to 14 of a 21-day cycle.

Arm B: Patients on the docetaxel arm received 60mg/m2 docetaxel as a 10-minute intravenous infusion on day 1 of a 21-day cycle and 8mg/10mg/12mg anlotinib orally daily on day 1to 14 of a 21-day cycle.

Approximately 18 patients will be enrolled to ensure that roughly 9 patients per arm complete treatments for primary endpoint analysis.

ELIGIBILITY:
Inclusion Criteria:

* Be≥18 years of age on the day of signing informed consent.
* Patients with histologic or cytologic confirmation of advanced or metastatic NSCLC with stage III or IV disease amenable to platinum-based chemotherapy were assessed for eligibility.
* Patients with EGFR、ALK、ROS1 Mutation-negative were eligible.
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Status.
* Life expectancy ≥3 months.
* Without serious system dysfunction and could tolerate chemotherapy.
* With normal marrow, liver ,renal and coagulation function:

a leucopenia count of ≥3.0×109/L; a platelet count of ≥1.5×109/L; hemoglobin≥ 90 g/L; a platelet count of ≥100×109/L; a alanine aminotransferase (ALAT) and aspartate aminotransferase (ASAT) of ≤2.5 UNL in case of liver metastasis; a total bilirubin (TBil) of ≤1.5 upper normal limitation (UNL); a creatinine (Cr) of ≤ 1.5 UNL; a creatinine clearance rate ≥ 50ml/min (Cockcroft-Gault);

* With normal coagulation function: activated partial thromboplastin time (APTT), prothrombin time (PT) and INR, each ≤ 1.5 x UNL.
* Female subjects of child-bearing potential must agree to use contraceptive measures starting 1 week before the administration of the first dose of apatinib until 8 weeks after discontinuing study drug. Male subjects must agree to use contraceptive measures during the study and 8 weeks after last dose of study drug.
* With written informed consent signed voluntarily by patients themselves or their supervisors witted by doctors.
* With good compliance and agree to accept follow-up of disease progression and adverse events.

Exclusion Criteria:

* Small cell lung cancer (include Small cell lung cancer mixture of NSCLC).
* Patients with brain or central nervous system metastases, including leptomeningeal disease, or CT/MRI examination revealed brain or leptomeningeal disease） (14 days before the random treatment has been completed and the symptoms of patients with brain metastases from stable can into the group, but need to the cerebral MRI, CT or vein angiography confirmed as without symptoms of cerebral hemorrhage).
* Iconography (CT or MRI) shows that the tumor vessels have 5 mm or less, or Cardiovascular involvement by Central tumor ; Or obvious lung empty or necrotic tumor.
* Uncontrollable hypertensive (systolic blood pressure or greater 140 mmHg or diastolic blood pressure or greater 90 mmHg, despite the best drug treatment).
* Significant cardiac disease as defined as: grade II or greater myocardial infarction, unstable arrhythmia(Including corrected QT interval (QTc )period between male or greater 450 ms, female or greater 470 ms); New York Heart Association (NYHA) grade II or greater heart dysfunction , or Echocardiography reveal left ventricular ejection fraction （LVEF）Less than 50%.
* Abnormal coagulation (INR > 1.5 or prothrombin time (PT) > ULN + 4 seconds or APTT ULN > 1.5), with bleeding tendency or be treated with thrombolysis and anticoagulation.

Note: under the premise of International Normalized ratio (INR) of prothrombin time (PT) Less than or equal to 1.5, allow to administrate low-dose heparin (adult daily dose is 06000 ~ 12000 U) or low-dose aspirin (100 mg daily dosage or less) , for prophylactic purposes.

* Urine routines show urine protein≥ ++, or urine protein quantity≥ 1.0 g during 24 hours.
* Patients with NCI-CTCAE grade II or greater peripheral neuropathy, except due to trauma.
* Clinically significant serous effusion (including pleural effusion, ascites, pericardial effusion).
* Serious, non-healing wound, ulcer, or bone fracture.
* Patients with severe infections , and need to receive Systemic antibiotic treatment.
* Decompensated diabetes or high dose glucocorticoid treatment of other contraindication.
* Active or chronic hepatitis c and/or Hepatitis B virus (HBV) infection.
* Has an obvious factor influencing oral drug absorption, such as unable to swallow, chronic diarrhea and intestinal obstruction, etc.
* Has received major surgery or severe traumatic injury, fractures or ulcer Within 4weeks before Random.
* Severe weight loss (> 10%) Within 6 weeks before Random.
* Has Clinically significant hemoptysis Within 3 months before Random (daily hemoptysis than 50 ml;Or significant clinical significance of bleeding symptoms or have definite bleeding tendency, such as gastrointestinal bleeding, bleeding ulcers, baseline period + + and above of fecal occult blood, or vasculitis, etc.
* Has venous thromboembolism events Within 12 months before Random, such as cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism, etc.
* There are any contraindications with receiving pemetrexed or docetaxel treatment; has a history of severe allergic reactions of docetaxel or other containing Polysorbate 80 (twain 80)
* There are allergic reaction to contrast media, anlotinib, and/or excipient of experimental drug.
* Patients with any other medical condition or reason, in that investigator's opinion, makes the patient unstable to participate in a clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2018-07-01 (Estimated); Primary Completion 2018-09-01 (Estimated); Study Completion 2018-10-01 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity | From enrollment to completion of study. Estimated about 6 months.
  Dose Limiting Toxicity (DLT) is referred to grade 3 non-hematological toxicity or grade 4 hematological toxicity according to NCI CTCAE 4.03 criteria
Maximum tolerance dose | From enrollment to completion of study. Estimated about 6 months
  Maximum Tolerance Dose (MTD) is the dose of treatment in the cohort where there are 2 cases of DTL reported.

SECONDARY OUTCOMES:
disease control rate | From enrollment to 2 months after treatment
  Clinical response of treatment according to RESIST v1.1 criteria (DCR, disease control rate)
time to progression | From enrollment to progression of disease. Estimated about 6 months.
  The length of time from enrollment until the time of progression of disease (TTP, time to progression).

CONTACTS AND LOCATIONS:
Overall Officials: Lin Gen, Principal Investigator — Fujian Cancer Hospital